CLINICAL TRIAL: NCT00347386
Title: Zinc as an Immunomodulator in the Treatment of Possible Serious Bacterial Infections in Infants 7 Days and up to 4 Months of Age
Brief Title: Therapeutic Zinc in Infant Bacterial Illness
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre For International Health (Other)
Collaborators: All India Institute of Medical Sciences (Other)
Responsible Party: Tor A Strand/ Researcher, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCO-CT-2004-003740-3
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Sepsis; Bacterial Infections; Pneumonia
Keywords: Infants; India; Zinc; Bacterial illness; Treatment
MeSH Terms: conditions — Sepsis; Bacterial Infections; Pneumonia | interventions — Zinc; Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zinc (Experimental): Administration of zinc sulphate every day during illness
  Interventions: Drug: Drug: Zinc (zinc sulphate)
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drug: Zinc (zinc sulphate) — Dissolvable tablet 10 mg. Once daily during the illness
  Other Names: Produced by Nutriset; Malaunay, France
  Arms: Zinc
Drug: Placebo — Placebo tablet, once daily
  Other Names: Produced by Nutriset; Malaunay, France
  Arms: Placebo

SUMMARY:
Infections are the important cause of high mortality in young infants in developing countries. Zinc is a crucial micronutrient as it influences various immune mechanisms and modulates host resistance to several pathogens. It has shown benefits as an adjunct therapy in infections like diarrhea and pneumonia in older children Given the predisposition of young infants in developing countries to zinc deficiency and infections, addition of zinc to standard treatment of serious bacterial infections may lead to significant improvements in the outcomes.

Several hypotheses will be examined in this clinical trial. The primary objective is to measure, in a double blind randomized controlled trial, the efficacy of giving 2 RDA (Required Daily Allowance 10 mg) of zinc orally in addition to routine antibiotics, for treatment of possible serious bacterial infection in infants >= 7 days and up to 4 months of age in reducing the proportion of treatment failures and time to discharge from the hospital. This will evaluate the clinical consequences of the possible immunomodulation by zinc supplementation. This is critical to demonstrate because nearly 80% of infant mortality occurs in first months of life.

Young infants with possible serious bacterial infections fulfilling the inclusion criteria will be enrolled in the study and stratified into 4 groups on basis of weight for age 'z' scores < -2 z and >=- 2 z and whether he/she has diarrhea or not. Within each stratum the subjects will be randomized to receive zinc or placebo. Treatment failures will be defined by the need for a change of initial antibiotic therapy. The minimum duration of monitoring will be till clinical recovery (using predetermined criteria). Serum copper, serum ferritin and serum transferrin receptors will be determined at enrollment, 72 hours after enrollment and at discharge from the hospital. Concentrations of CRP and procalcitonin will be measured at baseline, 72 hours after enrolment and at clinical recovery.

Documentation of efficacy of addition of zinc to standard therapy may provide a simple and low-cost strategy to improve survival in serious infections in young infants. This is likely to have a significant impact on infant morbidity and mortality. It will be good example of using a simple immunomodulator beneficially in improving child health.

DETAILED DESCRIPTION:
Infant mortality rate continues to be high in most developing countries despite advances in child health care. Infections are the most important cause of deaths in infants. There is increasing recognition that nutritional deficiencies including micronutrients are important determinants of infection and their outcomes. Zinc is a crucial micronutrient as it influences various immune mechanisms and modulates host resistance to several pathogens. Supplementation with zinc has been documented to provide protection against common childhood infections. It has also shown benefits as an adjunct therapy in infections like diarrhea and pneumonia in older children. Given the predisposition of young infants in developing countries to zinc deficiency and infections, addition of zinc to standard treatment of serious bacterial infections may lead to significant improvements in the outcomes. This is critical to demonstrate because nearly 80% of infant mortality occurs in first 2 months of life.

The infant mortality rates in India continue to be in excess of 60 per 1000 live births. Neonatal mortality contributes to over 64% of the infant deaths particularly in those who are born low birth weight. Most of the other deaths occur in the second and third months. Serious systemic infections like sepsis and pneumonia constitute 30-40% of the causes of mortality. Any health programme that aims at reducing infant mortality rate needs to address mortality in the first two months of life.

Almost 90% of all low birth weight (LBW) babies are born in developing countries, particularly in the Indian subcontinent. Nearly 70% of these are small for gestational age unlike in the developed world where the bulk of low birth weight babies are preterms. Zinc deficiency during fetal development is documented to cause intra-uterine growth retardation and also impaired postnatal immune functions making these babies more susceptible to severe infections. Studies have shown good correlation between cord blood zinc, maternal zinc concentration and birth weights.

The zinc content of the breast milk decreases rapidly after birth. In addition, the requirements are likely to be high as young infants in developing countries live in high microbial load environment and are exposed to recurrent infections. Further, malnourished infants need more zinc for catch up growth. All these predispose them to develop zinc deficiency and infections. In a population based study by our group last year, nearly 40% of young infants had low plasma zinc despite being breast-fed, probably a reflection of inadequate tissue stores (unpublished data).

Zinc influences many aspects of the immune system starting with its effects on the barrier and various components of innate and acquired immunity. There is sufficient data from animal and human studies of increased host susceptibility to infections with zinc deficiency. A vicious cycle of infection and zinc deficiency exists. Infection reduces the plasma zinc concentration, which reflects the severity of the infection and inflammation. This may be observed early during the illness. Organs such as the skin, thymus, bones and the epithelium also become depleted during this process. Severe bacterial illnesses also lead to zinc redistribution. It is plausible that this redistribution increases the infection severity.

There is limited data on therapeutic effect of zinc supplementation on severe infections in young infants less than 4 months of age. A short inexpensive course of zinc for patients with serious bacterial infections can become a simple but potent intervention to reduce young infant mortality and morbidity. While the effects of zinc deficiency and of supplementation are reasonably well documented eventually the benefits on clinical outcome alone can result in its application.

ELIGIBILITY:
Inclusion Criteria:

Evidence of possible serious bacterial infection, defined as a CRP >= 12 mg/L and any one of the following clinical features:

Fever (axillary temperature >= 37.5 degrees C) or hypothermia (axillary temperature <35.5 degrees C).

Lethargic or unconscious. No attachment to the breast in breast fed infants. No suckling in breast fed infants. Convulsions in the present episode. Bulging fontanel.

* History of acute refusal of feed in the present episode.
* Acute history of excessive cry or irritability in the present episode.
* Fast breathing defined as >= 60 breaths/minute (on second count) for infants < 2 months and >= 50 breaths/min in infants 2 months up to 4 months.
* Grunting in the absence of any non infective cause.
* Cyanosis in the absence of any non infective cause.
* Severe chest in drawing.
* Unexplained shock.
* Diarrhea in present episode.

Exclusion Criteria:

* Congenital malformations e.g. hydrocephalus, structural CNS malformation.
* Severe birth asphyxia defined as:

  * One minute APGAR (if available) of < 4/10.
  * CT scan or MRI or EEG abnormalities if available suggestive of hypoxic ischemic encephalopathy.
* Known structural defects, which interfere with feeding, e.g.cleft palate esophageal abnormalities, intestinal atresia and stenosis, malrotation of the gut,anorectal malformation.
* Subjects requiring ventilation or ionotropic support.
* History of diarrhea in the present episode.
* Known inborn error of metabolism.
* Chronic disorders of other organs e.g. neonatal cholestasis, chronic renal failure, pre-existing seizure disorder.
* Infants born of known HIV mothers.
* Clinical suspicion of necrotising enterocolitis.
* Congenital heart disease.
* Any CVS malformation:

  * Congenital heart disease.
  * Cyanosis before present episode.
  * Presence of murmur > grade 3/6.
* Ambiguous genitalia.
* Known chromosomal abnormality.
* Infants requiring exchange transfusion.

Ages: 1 Week to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Actual)
Dates: Start 2005-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
proportion with treatment failures | Within 3 weeks after enrollment

SECONDARY OUTCOMES:
the effect of zinc administration on plasma zinc and copper | up to three weeks
The efficacy of zinc on the duration of severe bacterial illness | 3 weeks
The efficacy of zinc given during severe bacterial illness on markers of inflammation | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shinjini Bhatnagar, DNB, PhD, Principal Investigator — All India Institute of Medical Sciences
Locations (3):
- India (3):
  - Deen Dayal Upadhyay Hospital,, New Delhi, New Delhi
  - All India Institute Of Medical Sciences, New Delhi, New Delhi
  - Kalawati Saran Children Hospital, New Delhi, New Delhi

REFERENCES:
- [Background] Mahalanabis D, Bhan MK. Micronutrients as adjunct therapy of acute illness in children: impact on the episode outcome and policy implications of current findings. Br J Nutr. 2001 May;85 Suppl 2:S151-8. doi: 10.1079/bjn2000308. PMID 11509104
- [Background] Shankar AH, Prasad AS. Zinc and immune function: the biological basis of altered resistance to infection. Am J Clin Nutr. 1998 Aug;68(2 Suppl):447S-463S. doi: 10.1093/ajcn/68.2.447S. PMID 9701160
- [Background] Bhutta ZA, Bird SM, Black RE, Brown KH, Gardner JM, Hidayat A, Khatun F, Martorell R, Ninh NX, Penny ME, Rosado JL, Roy SK, Ruel M, Sazawal S, Shankar A. Therapeutic effects of oral zinc in acute and persistent diarrhea in children in developing countries: pooled analysis of randomized controlled trials. Am J Clin Nutr. 2000 Dec;72(6):1516-22. doi: 10.1093/ajcn/72.6.1516. PMID 11101480
- [Background] Bhutta ZA, Black RE, Brown KH, Gardner JM, Gore S, Hidayat A, Khatun F, Martorell R, Ninh NX, Penny ME, Rosado JL, Roy SK, Ruel M, Sazawal S, Shankar A. Prevention of diarrhea and pneumonia by zinc supplementation in children in developing countries: pooled analysis of randomized controlled trials. Zinc Investigators' Collaborative Group. J Pediatr. 1999 Dec;135(6):689-97. doi: 10.1016/s0022-3476(99)70086-7. PMID 10586170
- [Background] Murray CJ, Lopez AD. Global mortality, disability, and the contribution of risk factors: Global Burden of Disease Study. Lancet. 1997 May 17;349(9063):1436-42. doi: 10.1016/S0140-6736(96)07495-8. PMID 9164317
- [Background] UNICEF. The State of the Worlds Children. New York, NY: Oxford University Press; 1999.
- [Background] Singh PP, Khushlani K, Veerwal PC, Gupta RC. Maternal hypozincemia and low-birth-weight infants. Clin Chem. 1987 Oct;33(10):1950. No abstract available. PMID 3665076
- [Background] Goel R, Misra PK. Study of plasma zinc in neonates and their mothers. Indian Pediatr. 1982 Jul;19(7):611-4. No abstract available. PMID 7174090
- [Background] Jeswani RM, Vani SN. A study of serum zinc levels in cord blood of neonates and their mothers. Indian J Pediatr. 1991 Sep-Oct;58(5):683-6. doi: 10.1007/BF02820191. PMID 1813415
- [Background] Prasad AS. Effects of zinc deficiency on Th1 and Th2 cytokine shifts. J Infect Dis. 2000 Sep;182 Suppl 1:S62-8. doi: 10.1086/315916. PMID 10944485
- [Background] Brown KH, Peerson JM, Rivera J, Allen LH. Effect of supplemental zinc on the growth and serum zinc concentrations of prepubertal children: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2002 Jun;75(6):1062-71. doi: 10.1093/ajcn/75.6.1062. PMID 12036814
- [Background] Cousins RJ, Leinart AS. Tissue-specific regulation of zinc metabolism and metallothionein genes by interleukin 1. FASEB J. 1988 Oct;2(13):2884-90. doi: 10.1096/fasebj.2.13.2458983.
- [Background] Zlotkin S, Arthur P, Schauer C, Antwi KY, Yeung G, Piekarz A. Home-fortification with iron and zinc sprinkles or iron sprinkles alone successfully treats anemia in infants and young children. J Nutr. 2003 Apr;133(4):1075-80. doi: 10.1093/jn/133.4.1075. PMID 12672922
- [Background] Dijkhuizen MA, Wieringa FT, West CE, Martuti S, Muhilal. Effects of iron and zinc supplementation in Indonesian infants on micronutrient status and growth. J Nutr. 2001 Nov;131(11):2860-5. doi: 10.1093/jn/131.11.2860. PMID 11694609
- [Background] Herman S, Griffin IJ, Suwarti S, Ernawati F, Permaesih D, Pambudi D, Abrams SA. Cofortification of iron-fortified flour with zinc sulfate, but not zinc oxide, decreases iron absorption in Indonesian children. Am J Clin Nutr. 2002 Oct;76(4):813-7. doi: 10.1093/ajcn/76.4.813. PMID 12324295
- [Background] Lind T, Lonnerdal B, Stenlund H, Ismail D, Seswandhana R, Ekstrom EC, Persson LA. A community-based randomized controlled trial of iron and zinc supplementation in Indonesian infants: interactions between iron and zinc. Am J Clin Nutr. 2003 Apr;77(4):883-90. doi: 10.1093/ajcn/77.4.883. PMID 12663287
- [Background] Schultink, W., Merzenich, M, Gross, R, Shrimpton, R, Dillon, D(1997). "Effects of iron-zinc supplementation on the iron, zinc, and vitamin A status of anamemic pre-school children. " Food and Nutrition Bulletin 18(4):311-16
- [Background] Abdulla M, Suck C. Blood levels of copper, iron, zinc, and lead in adults in India and Pakistan and the effect of oral zinc supplementation for six weeks. Biol Trace Elem Res. 1998 Mar;61(3):323-31. doi: 10.1007/BF02789092. PMID 9533570
- [Background] Brooks WA, Santosham M, Naheed A, Goswami D, Wahed MA, Diener-West M, Faruque AS, Black RE. Effect of weekly zinc supplements on incidence of pneumonia and diarrhoea in children younger than 2 years in an urban, low-income population in Bangladesh: randomised controlled trial. Lancet. 2005 Sep 17-23;366(9490):999-1004. doi: 10.1016/S0140-6736(05)67109-7. PMID 16168782
- [Background] Brooks WA, Yunus M, Santosham M, Wahed MA, Nahar K, Yeasmin S, Black RE. Zinc for severe pneumonia in very young children: double-blind placebo-controlled trial. Lancet. 2004 May 22;363(9422):1683-8. doi: 10.1016/S0140-6736(04)16252-1. PMID 15158629
- [Background] Bhandari N, Bahl R, Taneja S, Strand T, Molbak K, Ulvik RJ, Sommerfelt H, Bhan MK. Substantial reduction in severe diarrheal morbidity by daily zinc supplementation in young north Indian children. Pediatrics. 2002 Jun;109(6):e86. doi: 10.1542/peds.109.6.e86. PMID 12042580
- [Background] Strand TA, Chandyo RK, Bahl R, Sharma PR, Adhikari RK, Bhandari N, Ulvik RJ, Molbak K, Bhan MK, Sommerfelt H. Effectiveness and efficacy of zinc for the treatment of acute diarrhea in young children. Pediatrics. 2002 May;109(5):898-903. doi: 10.1542/peds.109.5.898. PMID 11986453
- [Derived] Singh P, Wadhwa N, Lodha R, Sommerfelt H, Aneja S, Natchu UC, Chandra J, Rath B, Sharma VK, Kumari M, Saini S, Kabra SK, Bhatnagar S, Strand TA. Predictors of time to recovery in infants with probable serious bacterial infection. PLoS One. 2015 Apr 24;10(4):e0124594. doi: 10.1371/journal.pone.0124594. eCollection 2015. PMID 25909192
- [Derived] Bhatnagar S, Wadhwa N, Aneja S, Lodha R, Kabra SK, Natchu UC, Sommerfelt H, Dutta AK, Chandra J, Rath B, Sharma M, Sharma VK, Kumari M, Strand TA. Zinc as adjunct treatment in infants aged between 7 and 120 days with probable serious bacterial infection: a randomised, double-blind, placebo-controlled trial. Lancet. 2012 Jun 2;379(9831):2072-8. doi: 10.1016/S0140-6736(12)60477-2. PMID 22656335